CLINICAL TRIAL: NCT05706610
Title: A Pilot Feasibility Trial of a Tailored Intervention to Improve Adherence in Adolescents and Young Adults With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: St. Jude Children's Research Hospital (Other); Seattle Children's Hospital (Other); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21CA268945 (NIH)
Record Dates: First submitted 2023-01-11; First posted 2023-01-31 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Cancer; Adherence, Medication
Keywords: cancer; adherence
MeSH Terms: conditions — Neoplasms; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored Program (Experimental): 8-week tailored program including 4 coach visits and 4 bi-weekly text check-ins
  Interventions: Behavioral: Tailored Program
- Feedback Program (Other): 8-week feedback program including 8 weekly texts
  Interventions: Behavioral: Feedback Program

INTERVENTIONS:
Behavioral: Tailored Program — Participants in the tailored program will participate in 4 sessions with a coach, 1 every other week. During these sessions, the AYA will work with their coach to identify a barrier to adherence to target and create an action plan using evidence-based behavior change techniques to address this barrier. In between sessions (on alternating weeks), the coach will check-in with a text including a reminder about the action plan and a calendar of the AYA's eCAP adherence data.
  Arms: Tailored Program
Behavioral: Feedback Program — Participants in the Feedback Program will receive weekly text messages including: a calendar depicting their weekly adherence (per eCAP data) and guidance for requesting additional support as desired.
  Arms: Feedback Program

SUMMARY:
A pilot feasibility randomized clinical trial comparing a tailored intervention to uniform standard of care will be conducted. A total of 40 AYAs with cancer will be randomized to one of the two programs. Data will be collected to explore the hypotheses that the intervention meets pre-established enrollment, retention, fidelity, and data completion feasibility criteria and that AYAs will rate the intervention as easy to use and acceptable.

DETAILED DESCRIPTION:
The proposed research includes a randomized clinical trial of a tailored adherence-promotion intervention (Tailored Program) as compared to uniform standard of care (Feedback Program) for adolescents and young adults with cancer. Up to 40 adolescents and young adults (AYAs) with cancer will be enrolled in this study. Participants who enroll in this trial will be given an eCAP electronic monitor, a pill bottle with a computer chip in the cap, to store their medication. After using the electronic monitor for 4 weeks to assess baseline adherence, participants who demonstrate non-adherence and have used the electronic monitor without difficulty will be asked to complete pre-treatment questionnaires. Next, participants will be randomly assigned to either the tailored adherence-promotion intervention group (Tailored Program) or the uniform standard of care group (Feedback Program). Participants will be assigned in a 1:1 ratio so that, at the end of the study, an equal number of participants will have been randomized to each group.

Participants in the tailored program will participate in 4 sessions with a coach, 1 every other week. During these sessions, the AYA will work with their coach to identify a barrier to adherence to target and create an action plan using evidence-based behavior change techniques to address this barrier. In between sessions (on alternating weeks), the coach will check-in with a text including a reminder about the action plan and a calendar of the AYA's eCAP adherence data. Participants in the Feedback Program will receive weekly text messages including: a calendar depicting their weekly adherence (per eCAP data) and guidance for requesting additional support as desired.

Adolescents and young adults will continue to use the electronic monitor to store their medication until approximately a month after their program ends. After their program ends, participants will complete post-treatment questionnaires regarding program usability and acceptability as well as their adherence.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 15 and 24 years of age
* Patient diagnosis of cancer
* Patient prescribed oral chemotherapy or prophylactic medication

Exclusion Criteria:

* Patient is not fluent in English
* Patient evidences significant cognitive deficits per medical team
* Patient's medical status or treatment precludes participation per medical team, patient, or caregiver
* Patient demonstrates greater than or equal to 95% adherence during run-in period
* Patient declines to use electronic monitoring device

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meghan E McGrady, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (3):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McGrady ME, Ketterl TG, Webster RT, Burns MMK, Bills SE, Burke M, Szulczewski L, Brock MY, Schwartz LE, Herriott JK, Hommel KA, Pai ALH, Mara CA, Norris RE. Feasibility Trial of a Tailored Adherence-Promotion Intervention for Adolescents and Young Adults With Cancer. Pediatr Blood Cancer. 2026 Jan;73(1):e32127. doi: 10.1002/pbc.32127. Epub 2025 Oct 27. PMID 41146444
- [Derived] McGrady ME, Ketterl TG, Webster RT, Schwartz LE, Brock MY, Szulczewski L, Burke M, Hommel KA, Pai ALH, Mara CA, Steele AC, Regan GG, Norris RE. Feasibility pilot trial of a tailored medication adherence-promotion intervention for adolescents and young adults with cancer: Study design and protocol. Contemp Clin Trials. 2024 Apr;139:107483. doi: 10.1016/j.cct.2024.107483. Epub 2024 Feb 29. PMID 38431133

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 70 enrolled participants, 24 met inclusion criteria and were randomized to one of the two intervention conditions
Period: Overall Study
Arm/Group | Tailored Program | Feedback Program
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tailored Program | Feedback Program | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.25 (2.47) | 18.73 (2.50) | 18.99 (2.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 0 | 1
  More the one race | 0 | 1 | 1
  Other race | 1 | 0 | 1
  White | 9 | 10 | 19
  I don't know | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Enrollment Rate
Description: Percent of approached eligible participants enrolling in the study
Time Frame: End of study enrollment period, approximately 12 months after enrollment initiation
Measure: Count of Participants; unit: Participants
Groups:
- Overall: Enrollment and retention were calculated at the study level
Arm/Group | Overall
Number analyzed (Participants) | 77
Participants | 70

2. Secondary Outcome: Retention Rate
Description: The percent of participants completing all procedures for which they were eligible The numerator is calculated via the following formula: (n AYAs eligible to complete at least some study procedures [n enrolled AYAs - n AYAs meeting criteria for unenrollment prior to study start] - n AYAs who never started study procedures - n AYAs who did not complete at least some study procedures) The denominator (n AYAs eligible to complete at least some study procedures) is calculated via the following formula: (n enrolled AYAs - n AYAs meeting criteria for unenrollment prior to study start)
Time Frame: From enrollment to study completion (approximately 4 weeks for patients deemed ineligible after run-in and approximately 16 weeks for patients deemed eligible after run-in)
Population: In all, 65 AYAs were eligible to complete at least some study procedures (70 enrolled - 5 meeting criteria for unenrollment prior to start = 65). Of these, 56 (65 - 8 AYAs who never started - 1 AYA who did not complete at least some study procedures = 56) completed all study procedures for which they were eligible, resulting in a retention rate of 86% (56/65).
Measure: Count of Participants; unit: Participants
Arm/Group | Overall
Number analyzed (Participants) | 65
Participants | 56

3. Secondary Outcome: Intervention Fidelity: Contact
Description: Percent of participants randomized to the Tailored Program who completed 4 intervention sessions
Time Frame: From randomization to the Tailored Program (at approximately week 4) to the completion of the Tailored Program (at approximately week 12) (total duration = approximately 8 weeks)
Population: This outcome is relevant to the Tailored Program only. Data from 2 participants who met criteria for unenrollment during the Tailored Program, and thus received fewer than 4 sessions due to no longer being eligible, are not included
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Program | Feedback Program
Number analyzed (Participants) | 10 | 0
Participants | 10 |

4. Secondary Outcome: Intervention Fidelity: Length
Description: Percent of participants randomized to the Tailored Program for whom all sessions were 30-45 minutes in length
Time Frame: as for outcome 3
Population: This outcome is relevant to the Tailored Program only.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Program | Feedback Program
Number analyzed (Participants) | 12 | 0
Participants | 8 |

5. Secondary Outcome: Intervention Fidelity: Duration
Description: Percent of randomized to the Tailored Program who completed all 4 intervention sessions during a 8-10 week period
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Program | Feedback Program
Number analyzed (Participants) | 10 | 0
Participants | 10 |

6. Secondary Outcome: Intervention Fidelity: Content
Description: Percent of participants randomized to the Tailored Program who received all of the planned intervention content as defined in the fidelity checklist
Time Frame: as for outcome 3
Population: This outcome is relevant to participants randomized to the tailored program only
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Program | Feedback Program
Number analyzed (Participants) | 12 | 0
Participants | 12 |

7. Secondary Outcome: Assessment Completion
Description: Percent of enrolled participants with complete data
Time Frame: From enrollment to the completion of post-intervention assessment which occurred approximately 4 weeks after program completion (total time frame = approximately 16 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Program | Feedback Program
Number analyzed (Participants) | 12 | 12
Participants | 12 | 12

8. Secondary Outcome: System Usability Scale
Description: A 10-item rating of usability, range = 0-100, better scores indicate better usability
Time Frame: Post-intervention assessment, approximately 4 weeks after program completion and approximately 16 weeks after enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored Program | Feedback Program
Number analyzed (Participants) | 12 | 12
score on a scale | 80.42 (13.05) | 81.25 (11.15)

9. Secondary Outcome: "Adjective Rating Scale" (Measure of Usability)
Description: 1-item rating of user friendliness, range = 1 (worst imaginable) to 7 (best imaginable), higher scores indicate better usability
Time Frame: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored Program | Feedback Program
Number analyzed (Participants) | 12 | 12
score on a scale | 5.92 (1.08) | 5.75 (0.97)

10. Secondary Outcome: Number of Participants Rating Behavioral Treatment Acceptability as 4 or Greater
Description: Rating of behavioral treatment acceptability - "I would recommend this program to other adolescents and young adults"; Possible range = 1 (strongly disagree) - 5 (strongly agree), better scores represent better acceptability; Dichotomous variable created representing whether participants scored this item as 1-3 (not acceptable) or 4-5 (acceptable)
Time Frame: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Program | Feedback Program
Number analyzed (Participants) | 12 | 12
Participants | 11 | 8

11. Secondary Outcome: Medical Adherence Measure
Description: 1-item self-report of missed doses
Time Frame: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage of doses taken
Arm/Group | Tailored Program | Feedback Program
Number analyzed (Participants) | 12 | 12
percentage of doses taken | 97.62 (5.56) | 90.28 (15.71)

12. Secondary Outcome: Electronically Monitored Medication Adherence
Description: Each participant will be given an electronic monitoring device to store their medication. The electronic monitoring device records each time the device is opened.
Time Frame: Starting 4 weeks prior to treatment initiation (approximately weeks 1-4) and continuing until 4 weeks after program completion (approximately weeks 12-16)
Population: Two participants had their medication discontinued prior to the end of the study period and thus do not have electronic adherence monitoring device data
Measure: Mean (Standard Deviation); unit: percentage of doses taken
Arm/Group | Tailored Program | Feedback Program
Number analyzed (Participants) | 10 | 12
percentage of doses taken | 85.44 (14.38) | 63.25 (30.84)

ADVERSE EVENTS:
Time Frame: 4 month study period
Description: Death obtained via electronic medical record review, other adverse events identified by participant report
Arm/Group | Tailored Program | Feedback Program
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT05706610/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/10/NCT05706610/ICF_000.pdf